CLINICAL TRIAL: NCT02159547
Title: Study of Comparing Dexketoprofen to Placebo in Migraine Attack
Brief Title: IV Dexketoprofen vs Placebo in Migranie Attack
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Cenker Eken, Associated Proffesor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 41/10
Record Dates: First submitted 2014-05-31; First posted 2014-06-10 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Migraine
Keywords: migraine, emergency department, dexketoprofen, placebo
MeSH Terms: conditions — Migraine Disorders; Emergencies | interventions — dexketoprofen trometamol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexketoprofen (Active Comparator): 50 mg intravenous dexketoprofen in 50 ml normal saline in 5 minutes infusion.
  Interventions: Drug: Dexketoprofen
- normal slaline (Placebo Comparator): 50 ml normal saline
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Dexketoprofen — 50 mg intravenous arveles in 50 ml saline in 5 minutes
  Other Names: Arveles
  Arms: Dexketoprofen
Other: Normal Saline — 50 ml normal saline
  Arms: normal slaline

SUMMARY:
H0 hypothesis: IV dexketoprofen is equivalent to placebo in ceasing migraine attack in emergency department.

H1 hypothesis: IV dexketoprofen is not equivalent (superior) to placebo in ceasing migraine attack in emergency department.

DETAILED DESCRIPTION:
Migraine attack is one of the most leading causes presentations to emergency department. Patients with migraine attack seek urgent care to cease their pain. There are so many interventions defined in the medical literature that can be used in migraine attacks. However, as a IV drug, dexketoprofen; little known whether IV dexketoprofen is superior to placebo or not. In the present study we aimed to determine the effects of IV dexketoprofen in migraine attack in emergency department.

ELIGIBILITY:
Inclusion Criteria:

* patients presented with headache who diagnosed as migraine attack according to the international headache society

Exclusion Criteria:

* denied to give inform concent, illiterate patients, chronic renal failure, taking NSAIDs during the last six hours, pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Gungor, Pyhsician, Principal Investigator — Antalya Training and Govermental Hospital
Locations (1):
- Antalya Training and Govermental Hospital, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Turkcuer I, Serinken M, Eken C, Yilmaz A, Akdag O, Uyan E, Kiray C, Elicabuk H. Intravenous paracetamol versus dexketoprofen in acute migraine attack in the emergency department: a randomised clinical trial. Emerg Med J. 2014 Mar;31(3):182-5. doi: 10.1136/emermed-2013-203044. Epub 2014 Jan 6. PMID 24394884

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexketoprofen | Normal Slaline
Started | 112 | 112
Completed | 112 | 112
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexketoprofen | Normal Slaline | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (11.1) | 37.6 (10.7) | 36.9 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 83 | 168
  Male | 27 | 29 | 56
Region of Enrollment [Number; unit: participants]
  Turkey | 112 | 112 | 224

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale Change
Description: Change from baseline in Visual Analogue Scale, 100 mm, at 45th minutes. Visual Analogue Scale is measurement tool scoring tool between 0 (no pain) and 100 mm (worst pain). Minimum clinically significant change in pain score is 13 or 16 mm.
Time Frame: 45 minutes
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Dexketoprofen | Normal Slaline
Number analyzed (Participants) | 112 | 112
units on a scale | 55 [49 to 60] | 30 [25 to 35]

2. Secondary Outcome: Adverse Effects
Description: The adverse effects is being recorded to the study form after the study drugs are administered at the 45th minutes.
Time Frame: 45th minutes
Measure: Number; unit: participants
Arm/Group | Dexketoprofen | Normal Slaline
Number analyzed (Participants) | 112 | 112
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dexketoprofen | Normal Slaline
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/112
Other Adverse Events (participants affected / at risk) | 0/112 | 0/112

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No